CLINICAL TRIAL: NCT05082753
Title: Randomized, Two-way, Two-period, Single Oral Dose, Open-label, Crossover, Bioequivalence Study to Compare Two Tablets of Ivermectin Tablets (3 mg Ivermectin) Versus Two Tablets of Stromectol ® Tablets (3 mg Ivermectin), in Healthy Subjects Under Fasting Conditions
Brief Title: Bioequivalence Study to Compare Two Tablets of Ivermectin Tablets (3 mg Ivermectin) Versus Two Tablets of Stromectol ® Tablets (3 mg Ivermectin), in Healthy Subjects Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 988-2020
Record Dates: First submitted 2021-09-13; First posted 2021-10-19 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Anthelmintic Agent
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ivermectin tablets (3 mg Ivermectin) (Experimental)
  Interventions: Drug: Ivermectin tablets (3 mg Ivermectin); Drug: Stromectol ® tablets
- Stromectol ® tablets (3 mg Ivermectin) (Active Comparator)
  Interventions: Drug: Ivermectin tablets (3 mg Ivermectin); Drug: Stromectol ® tablets

INTERVENTIONS:
Drug: Ivermectin tablets (3 mg Ivermectin) — Two Ivermectin tablets were administered orally.
Drug: Stromectol ® tablets — Two Ivermectin tablets were administered orally.

SUMMARY:
Randomized, two-way, two-period, single oral dose, open-label, crossover, bioequivalence study to compare two tablets of Ivermectin tablets (3 mg Ivermectin) versus two tablets of Stromectol ® tablets (3 mg Ivermectin), in healthy subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* The subject is aged between eighteen to fifty years (18 - 50), both inclusive.
* The subject is within the limits for his height & weight as defined by the body mass index range (18.5 - 30.0 Kg/m2).
* The subject is willing to undergo the necessary pre- & post- medical examinations set by this study.
* The results of medical history, physical examination, vital signs & conducted medical laboratory tests are normal as determined by the clinical investigator.
* The subject tested negative for hepatitis (B & C) viruses and human immunodeficiency virus (HIV).
* There is no evidence of psychiatric disorder, antagonistic personality, and poor motivation, emotional or intellectual problems likely to limit the validity of consent to participate in the study or limit the ability to comply with protocol requirements.
* The subject is able to understand and willing to sign the informed consent form.
* For female subjects: negative pregnancy test and the woman is using two reliable contraception methods
* The subject has normal cardiovascular system & ECG recording.
* The subject kidney functions test and liver enzymes (AST & ALT enzymes) are within normal range.

Exclusion Criteria:

* The subject is a heavy smoker (more than 10 cigarettes per day).
* The subject has suffered an acute illness one week before dosing.
* The subject has a history of or concurrent abuse of alcohol.
* The subject has a history of or concurrent abuse of illicit drugs.
* The subject has a history of hypersensitivity and/or contraindications to the study drug and any related compounds.
* The subject has been hospitalized within three months before the study or during the study.
* The subject is vegetarian.
* The subject has consumed caffeine or xanthine containing beverages or foodstuffs within two days before dosing and until 72 hours after dosing in all study periods.
* The subject has taken a prescription medication within two weeks or even an over the counter product (OTC) within one week before dosing in each study period and any time during the study, unless otherwise judged acceptable by the clinical investigator.
* The subject has taken grapefruit containing beverages or foodstuffs within seven (7) days before first dosing and any time during the study.
* The subject has been participating in any clinical study (e.g. pharmacokinetics, bioavailability and bioequivalence studies) within the last 80 days prior to the present study.
* The subject has donated blood within 80 days before first dosing.
* The subject has a history or presence of cardiovascular, pulmonary, renal, hepatic, gastrointestinal, hematological, endocrinal, immunological, dermatological, neurological, musculoskeletal or psychiatric diseases.
* The subject has consumed drugs or foodstuffs that may affect pharmacological or pharmacokinetic properties (for example: barbiturates (such as phenobarbital, butalbital), benzodiazepines (such as clonazepam, lorazepam), sodium oxybate (GHB), valproic acid, warfarin.) two weeks before dosing, during the study and two weeks after dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | 72 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for Cmax
AUC0-72 (due to Ivermectin long half-life) | 72 hours
  Statistical analysis of primary endpoints will include descriptive statistics, Analysis of Variance (ANOVA), and Confidence Interval (CI). The average bioequivalence of the products is concluded if the two-sided 90 % CI for the test to reference ratio of the population means is within 80.00 - 125.00 % for each of the Ln-transformed data for AUC0-72

SECONDARY OUTCOMES:
Tmax | 72 hours
  The descriptive statistics including Maximum, Minimum and Median values will be measured for Tmax
Blood pressure (safety and tolerability) | at pre-dosing; 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48 and 72 hours post-dosing, ±45 minutes of scheduled time
  Clinically significant abnormal deviations. Normal range of blood pressure > 90/60 and <140/90 mmHg.
Pulse (safety and tolerability) | at pre-dosing; 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 6, 8, 12, 24, 48 and 72 hours post-dosing, ±45 minutes of scheduled time
  Clinically significant abnormal deviations. Normal range of Pulse 60-100 b/m
Temperature (safety and tolerability) | at pre-dosing; 4, 12, 24, 48 and 72 hours post-dosing, ±45 minutes of scheduled time
  Clinically significant abnormal deviations. Normal range of temperature 36.5-37.5 ºC

CONTACTS AND LOCATIONS:
Overall Officials: Hakan Gürpınar, Study Director — Humanis Saglık
Locations (1):
- ACDIMA Biocenter, Amman, Jordan